CLINICAL TRIAL: NCT05121649
Title: Video Streaming in Norwegian Emergency Medical Call Centers as a Supplement to Telephone-instructed Bystander First Aid for Injured Patients
Brief Title: Video-instructed First Aid in Emergency Medical Call Centers
Status: Completed | Type: Observational
Sponsor: Oslo Metropolitan University (Other)
Collaborators: Vestre Viken Hospital Trust (Other); Laerdal Foundation (Other); Ostfold Hospital Trust (Other); Oslo University Hospital (Other); University Hospital of North Norway (Other); Helse Stavanger HF (Other Government)
Responsible Party: Principal Investigator, Magnus Hjortdahl, Associate professor, MD, Oslo Metropolitan University
Other Study IDs: 247264
Record Dates: First submitted 2021-10-25; First posted 2021-11-16 (Actual); Last update posted 2023-11-01 (Actual); Status verified 2023-10

CONDITIONS: Injuries; Emergencies
Keywords: emergency call center; dispatcher; video; first aid; emergency call
MeSH Terms: conditions — Wounds and Injuries; Emergencies

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Before: Injured patients included in the study from health trusts where video streaming not yet has been implemented in the EMCC
- After: Injured patients included in the study from health trusts where video streaming has been implemented in the EMCC
  Interventions: Other: Video streaming

INTERVENTIONS:
Other: Video streaming — Video streaming as a supplement to telephone during emergency calls for dispatchers at EMCCs
  Groups: After

SUMMARY:
Video streaming as an additional tool to telephone was introduced in some Norwegian emergency medical call centers during the spring of 2020. This allows the dispatchers to communicate with the caller through video streaming during emergency calls. Some studies are conducted on this use of video streaming, but further research is needed.

In this study, the investigators have chosen to focus on potential effect from video streaming on bystander first aid for injured patients. The investigators have knowledge from preliminary results that dispatchers often find video streaming useful in emergency calls regarding injuries.

This study will investigate whether the use of video streaming might have an effect on the recognition rate by dispatchers on the need for bystander first aid for injured patients. In addition, the investigators will investigate whether video-instructions from dispatcher can improve bystander first aid quality.

The investigators will be using data collected by ambulance personnel including patients with injuries, as well as data from EMCC journals and audio logs.

DETAILED DESCRIPTION:
Background:

Emergency Medical Communication Centres (EMCCs) in Norway receive more than 400 000 emergency calls every year, resulting in more than 250 000 ambulance dispatches. Emergency calls are answered by nurses or paramedics with special training, who by audio assesses the situation and decides on a response. Video streaming as a supplement to telephone in EMCC was introduced during springtime 2020 in Norway, and is independent of this study. The intended effect was to improve shared situational awareness between caller and operator, and thus improve the triage process. The video solution is live-only, and caller must give consent. Limited scientific evidence for such use exists, and even if video calls seems commonplace in society, the effects and acceptance in EMCCs has mainly been studied in simulated settings. Preliminary results from the early launch of video streaming showed that injured patients was one of the conditions where the dispatchers seemed to find video streaming useful. Previous studies by Bakke et.al investigating bystander first aid for injured patients, showed a potential for dispatchers in EMCCs to recognize more injured patients with the need for bystander first aid.

Aim:

This study focuses on the effect of video streaming in EMCCs on bystander first aid. The investigators aim to investigate whether dispatchers identifies the need for relevant first aid measures more frequently when using video streaming. The study will be conducted in several health trusts in Norway. In health trusts where video streaming not yet has been implemented in the EMCC, the investigators will collect data from period before video streaming is implemented, and after video streaming is implemented. From some health trusts in the study, video streaming already been implemented, and data collection will hence only be conducted for an after-period.

Methods and population size:

The number needed to treat is based on the studies by Bakke et al, as well it is based on one of our outcome goals: an aim for improvement of correctly identification of need for first aid by EMCC operator from 35% to 50%. Bakke et al included 355 cases during 18 months, which was done in a study area with approximately 270.500 inhabitants. For achievement of power of 0,80 and p-value <0,05 we need each study group to be 169, with the aimed improvement of 15%. Adding an estimate of missing cases of 10%, our study sample size for each group for this outcome measure is estimated to approximately 200 cases. For the outcome goal on quality improvement on first aid, which we aim the effect to be a raise in 20%, there is no aggregated outcome from previous studies to base an improvement on. The investigators therefore base our study sample size on number of cases included in Bakke's study. For this study to reach inclusion of 355 cases and with a study area with 1.150.000 inhabitants, the investigators need four months for each period. In Bakke's study, inclusion criteria were based on ICD-10 from hospital admissions. The investigators are therefore confident that the study will reach a minimum of 355 cases including patients not admitted to hospital as well. Based on these calculations on study sample sizes, the investigators estimate each of the before- and after periods to last 4 months, where cases before video implementation will be compared to calls after, separated by a wash-in period of 1-2 months.

Data collection and analyzes:

Patients will be included by ambulance personnel after the study's inclusion criteria. Ambulance personnel on scene will collect data through an internet-based questionnaire on need for first aid measures and quality of bystander first aid. In addition, data will be collected from EMCC journals and audio logs. This data will contain information on dispatchers recognition of first aid measures, as well as information on prehospital resources and time data. The investigators will also apply for data from the National Trauma Registry. Ambulance personnel participating in the data collection will complete an educational course about the questionnaire. The questionnaire used will be validated in a separate study. Analyzes of primary and secondary outcomes will be executed according to the ITT-principle. Uni- and multivariate regression analysis will be conducted.

Ethics:

The study is assessed by the Regional ethics committee in Norway as outside area of jurisdiction. It is approved by the Norwegian Center for Research Data and the Norwegian Health Directorate.

ELIGIBILITY:
Inclusion Criteria:

* Patient with an injury,
* One or more bystanders at scene,
* One or more of the following first aid measures have been attempted or should have been attempted: Open airway, bleeding control, recovery position, hypothermia prevention.

Exclusion Criteria:

* The caller is at a different location than the patient
* Patients who are alone on scene and contacted the EMCC themselves

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Patients with injuries who meet the inclusion criteria in the health trusts cooperating as study areas.
Sampling Method: Non-Probability Sample
Enrollment: 174 (Actual)
Dates: Start 2021-11-08 (Actual); Primary Completion 2023-02-28 (Actual); Study Completion 2023-06-30 (Actual)

PRIMARY OUTCOMES:
Dispatchers' recognition of relevant first aid measures | Through study completion, an average of 1,5 years
  Number of patients where dispatchers in the EMCCs recognizes relevant first aid measures

SECONDARY OUTCOMES:
First aid measures performed by bystander | Through study completion, an average of 1,5 years
  Number of patients with first aid measures performed by bystander before the arrival of the first ambulance unit
Bystander first aid quality | Through study completion, an average of 1,5 years
  Number of patients with first aid measures of high quality performed by bystander

OTHER OUTCOMES:
Time delay until activation of first ambulance | Through study completion, an average of 1,5 years
  No increase in time from the emergency call is received until activation of first ambulance unit
Time delay until need for first aid is recognized by dispatcher | Through study completion, an average of 1,5 years
  No increase in time from the emergency call is received until need for first aid is recognized by the dispatcher
30-days mortality for patients included | Through study completion, an average of 1,5 years
  No increase in 30-days mortality for patients where video streaming was used

CONTACTS AND LOCATIONS:
Overall Officials: Magnus Hjortdahl, PhD, Principal Investigator — OsloMet
Locations (1):
- University of OsloMet, Oslo, Norway

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bakke HK, Steinvik T, Ruud H, Wisborg T. Effect and accuracy of emergency dispatch telephone guidance to bystanders in trauma: post-hoc analysis of a prospective observational study. Scand J Trauma Resusc Emerg Med. 2017 Mar 7;25(1):27. doi: 10.1186/s13049-016-0343-z. PMID 28270170
- [Background] Ecker H, Lindacher F, Adams N, Hamacher S, Wingen S, Schier R, Bottiger BW, Wetsch WA. Video-assisted cardiopulmonary resuscitation via smartphone improves quality of resuscitation: A randomised controlled simulation trial. Eur J Anaesthesiol. 2020 Apr;37(4):294-302. doi: 10.1097/EJA.0000000000001177. PMID 32073408
- [Background] Lee JS, Jeon WC, Ahn JH, Cho YJ, Jung YS, Kim GW. The effect of a cellular-phone video demonstration to improve the quality of dispatcher-assisted chest compression-only cardiopulmonary resuscitation as compared with audio coaching. Resuscitation. 2011 Jan;82(1):64-8. doi: 10.1016/j.resuscitation.2010.09.467. Epub 2010 Oct 30. PMID 21036457
- [Background] Ecker H, Wingen S, Hamacher S, Lindacher F, Bottiger BW, Wetsch WA. Evaluation Of CPR Quality Via Smartphone With A Video Livestream - A Study In A Metropolitan Area. Prehosp Emerg Care. 2021 Jan-Feb;25(1):76-81. doi: 10.1080/10903127.2020.1734122. Epub 2020 Mar 20. PMID 32091293
- [Background] Lin YY, Chiang WC, Hsieh MJ, Sun JT, Chang YC, Ma MH. Quality of audio-assisted versus video-assisted dispatcher-instructed bystander cardiopulmonary resuscitation: A systematic review and meta-analysis. Resuscitation. 2018 Feb;123:77-85. doi: 10.1016/j.resuscitation.2017.12.010. Epub 2017 Dec 12. PMID 29242057
- [Background] Linderoth G, Lippert F, Ostergaard D, Ersboll AK, Meyhoff CS, Folke F, Christensen HC. Live video from bystanders' smartphones to medical dispatchers in real emergencies. BMC Emerg Med. 2021 Sep 6;21(1):101. doi: 10.1186/s12873-021-00493-5. PMID 34488626
- [Background] Bakke HK, Steinvik T, Eidissen SI, Gilbert M, Wisborg T. Bystander first aid in trauma - prevalence and quality: a prospective observational study. Acta Anaesthesiol Scand. 2015 Oct;59(9):1187-93. doi: 10.1111/aas.12561. Epub 2015 Jun 19. PMID 26088860
- [Background] Melbye S, Hotvedt M, Bolle SR. Mobile videoconferencing for enhanced emergency medical communication - a shot in the dark or a walk in the park? -- A simulation study. Scand J Trauma Resusc Emerg Med. 2014 Jun 2;22:35. doi: 10.1186/1757-7241-22-35. PMID 24887256
- [Background] Yang CW, Wang HC, Chiang WC, Hsu CW, Chang WT, Yen ZS, Ko PC, Ma MH, Chen SC, Chang SC. Interactive video instruction improves the quality of dispatcher-assisted chest compression-only cardiopulmonary resuscitation in simulated cardiac arrests. Crit Care Med. 2009 Feb;37(2):490-5. doi: 10.1097/CCM.0b013e31819573a5. PMID 19114904
- [Background] Bolle SR, Hasvold P, Henriksen E. Video calls from lay bystanders to dispatch centers - risk assessment of information security. BMC Health Serv Res. 2011 Sep 30;11:244. doi: 10.1186/1472-6963-11-244. PMID 21958387